CLINICAL TRIAL: NCT04750629
Title: Clinical Evaluation of a Point-of-Care (POC), SARS-CoV-2 CoviDx™ Rapid Antigen Test
Brief Title: Clinical Evaluation of a Point-of-Care (POC), COVID-19 Rapid Antigen Test (CoviDx™)
Acronym: CoviDx
Status: Completed | Type: Observational
Sponsor: Lumos Diagnostics (Industry)
Collaborators: Rapid Pathogen Screening (Industry)
Responsible Party: Sponsor
Other Study IDs: 21 0115
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: SARS-CoV-2; Covid19
Keywords: Antigen; Rapid; Point of care testing
MeSH Terms: conditions — COVID-19; Fasting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal Swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SARS-Cov-2 RT-PCR AND CoviDx Rapid Antigen Testing: Sequentially enrolled symptomatic patients who present for COVID-19 testing and have a swab collected for high-sensitive, SARS-CoV-2 RT-PCR testing per Standard of Care AND a swab for CoviDx™ Rapid Antigen testing.
  Interventions: Device: POC CoviDx™ Rapid Antigen Test

INTERVENTIONS:
Device: POC CoviDx™ Rapid Antigen Test — All patients will have a nasal swab for CoviDx™ Rapid Antigen testing

SUMMARY:
Prospective study that will evaluate the clinical agreement of the CoviDx™ Rapid Antigen test compared to SARS-CoV-2 RT-PCR.

DETAILED DESCRIPTION:
All patients who present with Covid-19-like symptoms within 5 days prior to consult, who consent to participate in the study, will undergo a nasopharyngeal swab (NP) collected for SARS-CoV-2 RT-PCR with EUA as per standard of care and nasal swab collection for CoviDx Rapid Antigen testing.

ELIGIBILITY:
Inclusion Criteria:

* Nasopharyngeal swab collected for SARS-CoV-2 RT-PCR with EUA as per standard of care within 3 hours of CoviDx Rapid Antigen Swab collection
* First onset of COVID-19-like symptoms within the last 5 days
* ≥ 1 year of age
* Signed Informed Consent

Exclusion Criteria:

* Unable or unwilling to provide signed, Informed Consent
* Less than 1 year of age
* SARS-Cov-2 RT-PCR collection that occurred > 3 hours from CoviDx Rapid Antigen Swab collection
* First onset of COVID-19-like symptoms occurring more than 5 days from study visit
* Invalid or missing PCR test results
* Use of a non-high-sensitive SARS-CoV-2 test as the qualifying SARS-CoV-2 RT-PCR test (e.g., Abbott ID NOW, rapid antigen tests, tests that do not have FDA EUA, a test that was not approved by Sponsor for use in the study)
* Enrollment in another study involving the collection of a nasopharyngeal or nasal swab
* Receipt of a COVID-19 vaccine or participation in a COVID-19 vaccine study

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Symptomatic patients who are suspected of having SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Sensitivity of SARS-CoV-2 antigen in nasal swab as compared to a high-sensitive SARS-CoV-2 RT-PCR granted Emergency Use Authorization (EUA) by the FDA | 30 days
  The primary outcome is the presence of SARS-CoV-2 antigen in nasal swab as compared to confirmatory diagnosis SARS-CoV-2 as determined by a high-sensitive SARS-CoV-2 RT-PCR granted Emergency Use Authorization (EUA) by the FDA

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Doral Medical Research, Hialeah, Florida
  - Comprehensive Clinical Research, West Palm Beach, Florida